CLINICAL TRIAL: NCT04936022
Title: Feasibility Study to Assess the Delivery of a Novel Isometric Exercise Intervention for People With Stage 1 Hypertension in the NHS
Brief Title: Isometric Exercise for People With Raised Blood Pressure
Acronym: IsoFIT-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Collaborators: University of Kent (Other); Canterbury Christ Church University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIHR200485; 13472393 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2021-04-19; First posted 2021-06-23 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
Keywords: Isometric exercise; Exercise; Hypertension; High blood pressure; General practice; Feasibility study
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Multi-centre randomized controlled feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): To receive standard care lifestyle advice only
  Interventions: Behavioral: Standard care lifestyle advice
- Isometric Exercise (Experimental): To receive standard care lifestyle advice plus 3 sessions of isometric exercise per week
  Interventions: Other: Isometric Exercise; Behavioral: Standard care lifestyle advice

INTERVENTIONS:
Other: Isometric Exercise — Prescribed 6 months of isometric exercise training (three sessions per week, comprised of 4 x 2-minute bouts with 2-minute recovery periods in-between).
  Arms: Isometric Exercise
Behavioral: Standard care lifestyle advice — Healthy lifestyle advice for hypertension, given by a healthcare professional.

SUMMARY:
High blood pressure affects many people in the United Kingdom. People with raised blood pressure (140-159/90-99 mmHg) are recommended to make changes in their lifestyle (e.g. smoking/alcohol/diet/exercise) and/or medication in order to reduce their blood pressure. Current knowledge suggests that a particular type of exercise - isometric exercise - can lower blood pressure. Isometric exercise involves holding a fixed body position for a short period of time. As most of the information about the benefits of this type of exercise comes from laboratory-based studies, researchers want to find out if it is possible for GP practices to offer NHS patients with clinically high blood pressure an isometric exercise plan to do at home and how it might affect their blood pressure over 6 months. They will also find out the experiences of those doing this type of exercise and whether it can be done consistently at home over time.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Clinic systolic BP 140-159 mmHg
* Able to provide informed consent

Exclusion Criteria:

* Currently taking anti-hypertensive medication
* White coat hypertension, as evidenced by averaged home systolic BP <135 mmHg
* Inability to undertake study intervention (isometric exercise)
* Previous history of any of the following:

  * Diabetes mellitus (Type 1 or type 2)
  * Ischaemic heart disease (myocardial infarction and/or coronary angina and/or coronary revascularization procedure)
  * Moderate or severe stenotic or regurgitant heart valve disease
  * Atrial or ventricular arrhythmia
  * Stroke or transient ischaemic attack
  * Aortic aneurysm and/or peripheral arterial disease
  * Uncorrected congenital or inherited heart condition
* Estimated glomerular filtration rate <45 ml/min (calculated using CKD-EPI or MDRD formulae, and taking most recent documented results)
* Documented left ventricular ejection fraction <45% and/or left ventricular hypertrophy (by either echocardiography or standard ECG criteria e.g. Sokolow-Lyon)
* Documented urine albumin:creatinine ratio >3.5 mg/mmol
* Inability to provide informed consent
* If female, pregnancy or currently breast feeding
* Enrolled in another Clinical Trial of an Interventional Medicinal Product or Medical Device or other interventional study
* Medical condition that, in the opinion of the investigator, would make the participant unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Experience of intervention delivery | Project month 11
  Qualitative focus groups with health care professionals identifying the type and number of each barrier and facilitator, of the practical delivery of isometric exercise intervention.
Change in systolic blood pressure (mmHg) from baseline to Week 4. | Participant week 4
Change in systolic blood pressure (mmHg) from baseline to Month 3. | Participant 3 months
Change in systolic blood pressure (mmHg) from baseline to Month 6. | Participant 6 months

SECONDARY OUTCOMES:
Early fidelity of the isometric exercise prescription. | Participant week 1
  Assessed by checking whether individual participant's heart rate (bpm) measures fall within 95% of their peak heart rate confidence intervals following the first three training sessions.
Short-term fidelity of the isometric exercise prescription. | Participant week 4
  Assessed by checking whether individual participant's heart rate (bpm) measures fall within 95% of their peak heart rate confidence intervals following the first four weeks (12) of training sessions.
Short-term adherence to the Isometric exercise (IE) training. | Participant week 4
  Measured using the proportion of participants (number) completing a minimum of 8 of 12 IE sessions up to the 4-week point.
Mid-term adherence to the Isometric exercise training. | Participant 3 Months
  Measured using the proportion of participants (number) completing a minimum of two thirds of all IE sessions up to 3 months.
Long-term adherence to the Isometric exercise training. | Participant 6 Months
  Measured using the proportion of participants (number) completing a minimum of two thirds of all IE sessions up to 6 months.
Recruitment rates from data collected at sites. | Project month 10
  This will be measured by calculating the average number of participants recruited per week.
Short-term attrition rates from data collected at sites. | Participant week 4
  This will be measured by calculating the number of withdrawals from the study up to 4 weeks.
Mid-term attrition rates from data collected at sites. | Participant 3 months
  This will be measured by calculating the number of withdrawals from the study up to 3 months.
Long-term attrition rates from data collected at sites. | Participant 6 months
  This will be measured by calculating the number of withdrawals from the study up to 6 months.
Change in diastolic blood pressure (mmHg) from baseline to Week 4. | Week 4
Change in diastolic blood pressure (mmHg) from baseline to Month 3. | Month 3
Change in diastolic blood pressure (mmHg) from baseline to Month 6. | Month 6
Experience of isometric exercise intervention. | Month 11
  Qualitative focus groups with study participants identifying the number of positive and negative experiences of the isometric exercise intervention and taking part in the study.
Participant experiences of undertaking isometric exercise. | Participant week 4.
  Collected using participant study-specific survey with closed and open questions.
Subjective opinion of healthcare professionals on their willingness to consider the intervention as a treatment option for patients with Stage 1 hypertension. | Project month 11.
  Collected using semi-structured interviews conducted by telephone with healthcare professionals from GP practices not taking part as study recruitment sites.
Short-term Quality-adjusted life years (QALYs) calculated from patients' responses to the EQ-5D-5L questionnaire. | Participant 4 weeks
  The health profile established from EQ-5D-5L will be converted into a utility index (0 and 1) using the validated mapping function to derive utility values for EQ-5D-5L from the existing EQ-5D-3L. These utilities will be multiplied by the time spent in each state to generate QALYs.
Mid-term Quality-adjusted life years calculated from patients' responses to the EQ-5D-5L questionnaire. | Participant 3 months
  The health profile established from EQ-5D-5L will be converted into a utility index (0 and 1) using the validated mapping function to derive utility values for EQ-5D-5L from the existing EQ-5D-3L. These utilities will be multiplied by the time spent in each state to generate QALYs.
Long-term Quality-adjusted life years calculated from patients' responses to the EQ-5D-5L questionnaire. | Participant 6 months
  The health profile established from EQ-5D-5L will be converted into a utility index (0 and 1) using the validated mapping function to derive utility values for EQ-5D-5L from the existing EQ-5D-3L. These utilities will be multiplied by the time spent in each state to generate QALYs.
Healthcare resource utilisation (a). | Participant 4 weeks.
  Measuring healthcare access by using the number of GP visits at 4 weeks.
Healthcare resource utilisation (a). | Participant 3 months
  Measuring healthcare access by using the number of GP visits at 3 months.
Healthcare resource utilisation (a). | Participant 6 months
  Measuring healthcare access by using the number of GP visits at 6 months.
Healthcare resource utilisation (b). | Participant 4 weeks.
  Measuring healthcare access by using the number of nurse visits at 4 weeks.
Healthcare resource utilisation (b). | Participant 3 months.
  Measuring healthcare access by using the number of nurse visits at 3 months.
Healthcare resource utilisation (b). | Participant 6 months.
  Measuring healthcare access by using the number of nurse visits at 6 months.
Healthcare resource utilisation (c). | Participant 4 weeks.
  Measuring healthcare access by using the number of other health professionals visits at 4 weeks.
Healthcare resource utilisation (c). | Participant 3 months.
  Measuring healthcare access by using the number of other health professionals visits at 3 months.
Healthcare resource utilisation (c). | Participant 6 months.
  Measuring healthcare access by using the number of other health professionals visits at 6 months.
Healthcare resource utilisation (d). | Participant 4 weeks.
  Measuring healthcare access by using the number of number of A&E attendances at 4 weeks.
Healthcare resource utilisation (d). | Participant 3 months.
  Measuring healthcare access by using the number of number of A&E attendances at 3 months.
Healthcare resource utilisation (d). | Participant 6 months.
  Measuring healthcare access by using the number of number of A&E attendances at 6 months.
Healthcare resource utilisation (e). | Participant 4 weeks.
  Measuring healthcare access by using the number of number of inpatient hospital admissions at 4 weeks.
Healthcare resource utilisation (e). | Participant 3 months.
  Measuring healthcare access by using the number of number of inpatient hospital admissions at 3 months.
Healthcare resource utilisation (e). | Participant 6 months.
  Measuring healthcare access by using the number of inpatient hospital admissions at 6 months.
Healthcare resource utilisation (f). | Participant 4 weeks.
  Measuring healthcare access by using the number of inpatient diagnostic tests at 4 weeks.
Healthcare resource utilisation (f). | Participant 3 months.
  Measuring healthcare access by using the number of inpatient diagnostic tests at 3 months.
Healthcare resource utilisation (f). | Participant 6 months.
  Measuring healthcare access by using the number of inpatient diagnostic tests at 6 months.
Intervention costs. | Participant 4 weeks.
  This will be measured by calculating the time cost of the training team and healthcare professionals, the cost of supplies and the equipment necessary to implement the intervention.
Intervention costs. | Participant 3 months.
  This will be measured by. calculating the time cost of the training team and healthcare professionals, the cost of supplies and the equipment necessary to implement the intervention.
Intervention costs | Participant 6 months.
  This will be measured by calculating the time cost of the training team and healthcare professionals, the cost of supplies and the equipment necessary to implement the intervention.
Medication at short-term time point (a) | Participant 4 weeks.
  Measured using the frequency per week in days, start and end date per medication at 4 weeks.
Medication at mid-term time point (a) | Participant 3 months.
  Measuring the frequency per week in days, start and end date per medication at 3 months.
Medication at long-term time point (a) | Participant 6 months.
  Measuring the frequency per week in days, start and end date per medication at 6 months.
Medication at short-term time point (b) | Participant 4 weeks.
  Measured using the dosage per day (mg), start and end date per medication at 4 weeks.
Medication at mid-term time point (b) | Participant 3 months.
  Measuring the dosage per day (mg), start and end date per medication at 3 months.
Medication at long-term time point (b) | Participant 6 months.
  Measuring the dosage per day (mg), start and end date per medication at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher K Farmer, Study Director — University of Kent
Locations (6):
- United Kingdom (6):
  - Canterbury Medical Practice, Canterbury, Kent
  - Kent and Canterbury Hospital, Canterbury, Kent
  - Newton Place Surgery, Faversham, Kent
  - St Helier Hospital, Carshalton, Surrey
  - Maywood Healthcare Centre, Bognor Regis, West Sussex
  - Brighton Health and Wellbeing Centre, Hove

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are/will be available upon request from Dr Jonathan Wiles (jim.wiles@canterbury.ac.uk). The data will become available 1 year after the study finishes which will be approximately December 2022 and may be accessed for up to 5 years. Anonymised data may be accessed by researchers at universities, NHS organisations or other healthcare providers where the sharing of data has a clearly defined purpose and its use will be of benefit to wider society. Data will be shared by secure data transfer. Consent from participants was obtained for the use of their information for future research and to be shared anonymously with other researchers.
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Wiles JD, Santer E, Rees-Roberts M, Borthwick R, Doulton T, Swift PA, Pellatt-Higgins T, Saxby K, Mills A, Gousia K, MacInnes D, O'Driscoll J, West A, Darby J, Short V, Farmer CK. Feasibility randomised controlled trial to assess the delivery of a novel isometric exercise intervention for people diagnosed with uncomplicated stage 1 hypertension in the National Health Service: key quantitative findings. BMJ Open. 2025 Jun 4;15(6):e091219. doi: 10.1136/bmjopen-2024-091219. PMID 40467325